CLINICAL TRIAL: NCT00744952
Title: VCRC Imaging Protocol for Magnetic Resonance and Positron Emission Tomography in Large-vessel Vasculitis (Takayasu's Arteritis):Development as Clinical Trial Outcome Measures
Brief Title: Use of MRI and PET for Assessing Disease Activity in Takayasu's Arteritis
Status: Completed | Type: Observational
Sponsor: Peter Merkel (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor-Investigator, Peter Merkel, Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Other Study IDs: VCRC5515; U54AR057319 (NIH)
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Takayasu Arteritis
Keywords: Large-vessel vasculitis
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Assessing disease activity in people with Takayasu's arteritis is difficult, as most people with the disease do not exhibit visible, measurable symptoms. Combination positron emission tomography/computed axial tomography (PET/CT) is a particularly sensitive, accurate scanning method that may improve researchers' ability to evaluate people with the disease. This study will determine the effectiveness of PET/CT in assessing disease activity in people with Takayasu's arteritis.

DETAILED DESCRIPTION:
Takayasu's arteritis is a rare inflammatory disease that affects the aorta and its branches. The disease is much more common in females than in males, and disease onset typically occurs between the ages of 15 and 30. People with this disease often experience general discomfort, fatigue, fever, night sweats, weight loss, and joint pain. In the late stages of the disease, weak arterial walls may lead to aneurysms. Many patients do not exhibit any visible symptoms until this point, however. Because many people with Takayasu's arteritis do not have overt disease symptoms, the assessment of disease activity is difficult. Laboratory tests can help, but are often unreliable. Novel approaches to assessing disease activity are urgently needed to enhance and facilitate research on Takayasu's arteritis. This study will determine the effectiveness of combination positron emission tomography/computed axial tomography (PET/CT) in assessing disease activity in people with Takayasu's arteritis.

Participants in this study will enroll while their disease is active. The first PET/CT scan will take place upon study entry, while there is active disease. Participants will have a second PET/CT scan 3 months later, and a third scan 3 months after that if there is still active disease present. Participants will have a maximum of 3 scans unless a scan needs to be repeated because of technical failures, though this does not often happen. If there is no active disease at the time of the second scan, a third scan will not be done. All PET/CT scans will be scheduled within 10 days of participants' routine MRI scans. This study will not require any follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Takayasu's arteritis, as defined by the VCRC Longitudinal Study #5503
* Currently enrolled in the VCRC Longitudinal Study #5503
* Active disease has occurred in conjunction with a disease relapse within 2 weeks before study entry (A detailed definition of "active disease" is available in the study protocol.)
* Willing and able to comply with the schedule for imaging studies and follow-up procedures

Exclusion Criteria:

* Pregnant or breastfeeding
* Unable to comply with study guidelines
* Unable to safely undergo MRI scanning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will have been diagnosed with Takayasu's arteritis and will be currently enrolled in the Vasculitis Clinical Research Consortium (VCRC) Longitudinal Study #5503.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Disease activity | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (5):
- United States (3):
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Toronto, Ontario

REFERENCES:
- [Background] Numano F. The story of Takayasu arteritis. Rheumatology (Oxford). 2002 Jan;41(1):103-6. doi: 10.1093/rheumatology/41.1.103. No abstract available. PMID 11792888
- [Background] Stone JH, Hoffman GS, Merkel PA, Min YI, Uhlfelder ML, Hellmann DB, Specks U, Allen NB, Davis JC, Spiera RF, Calabrese LH, Wigley FM, Maiden N, Valente RM, Niles JL, Fye KH, McCune JW, St Clair EW, Luqmani RA; International Network for the Study of the Systemic Vasculitides (INSSYS). A disease-specific activity index for Wegener's granulomatosis: modification of the Birmingham Vasculitis Activity Score. International Network for the Study of the Systemic Vasculitides (INSSYS). Arthritis Rheum. 2001 Apr;44(4):912-20. doi: 10.1002/1529-0131(200104)44:43.0.CO;2-5. PMID 11318006
- [Background] Weyand CM, Goronzy JJ. Medium- and large-vessel vasculitis. N Engl J Med. 2003 Jul 10;349(2):160-9. doi: 10.1056/NEJMra022694. No abstract available. PMID 12853590
- [Background] Tso E, Flamm SD, White RD, Schvartzman PR, Mascha E, Hoffman GS. Takayasu arteritis: utility and limitations of magnetic resonance imaging in diagnosis and treatment. Arthritis Rheum. 2002 Jun;46(6):1634-42. doi: 10.1002/art.10251. PMID 12115196
- [Background] Hoffman GS, Merkel PA, Brasington RD, Lenschow DJ, Liang P. Anti-tumor necrosis factor therapy in patients with difficult to treat Takayasu arteritis. Arthritis Rheum. 2004 Jul;50(7):2296-304. doi: 10.1002/art.20300. PMID 15248230
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/vcrc/